CLINICAL TRIAL: NCT05924282
Title: Impact of Positron-Emission-Tomography on the Surgical Treatment for Loco-regionally Recurrent Colorectal Cancer
Brief Title: PET on Surgery for Loco-regionally Recurrent Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202305096RINA
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: PET-driven Surgery; Loco-regional Recurrent Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sole PET group: Tumor recurrence was detected solely by PET; the surgery was performed and the extent of the resection was guided by the PET.
  Interventions: Procedure: Curative intent surgery
- Combined CT/MRI plus PET group: Tumor recurrence was detected by computed tomography (CT) / magnetic resonance imaging (MRI) and PET; the surgery was performed and the extent of the resection was guided by the CT/MRI+PET.
  Interventions: Procedure: Curative intent surgery
- Control group: Tumor recurrence was detected but no surgery was performed.

INTERVENTIONS:
Procedure: Curative intent surgery — Curative intent surgery means that surgeons intend to perform R0 resection.
  Groups: Combined CT/MRI plus PET group; Sole PET group

SUMMARY:
The influence of Positron-Emission-Tomography (PET) on the surgical treatment of loco-regionally recurrent colorectal cancer (LRRCRC) remains obscure and deserves further investigation.

DETAILED DESCRIPTION:
Loco-regionally recurrent colorectal cancer (LRRCRC) occurs in 4.0-11.5% of patients following treatment of primary colorectal cancer with curative intent, and can be categorized as peri-anastomotic, mesenteric/paracolic (nodal), retroperitoneal and peritoneal.1-4 In contrast to distant recurrences (e.g. liver, lung or bone metastasis), LRRCRCs is a less recognized clinical entity, although it is generally accepted that surgical resection remains the major treatment modality to provide the long-term survival for such patients.5-7 However, the value of resection for LRRCRC is obscure, given the role of surgical resection in treating LRRCRC has received comparatively little attention with a scant literature to draw upon when making treatment recommendations and no available consensus statements.8,9 Moreover, in clinical practice, it has been recognized that more than 50% of patients with recurrent colorectal cancer brought to the operating room for attempted curative surgery were unable to undergo the planned operation because more extensive disease than anticipated was discovered at laparotomy. Therefore, it has been suggested that a formal multidisciplinary team (MDT) discussion based on more precise diagnostic armamentariums be mandatory for more accurate evaluation of tumor burden and would allow curative surgery to be offered to a better-selected group of patients with recurrent colorectal malignancy10-14.

Remarkably, Positron-Emission-Tomography (PET) scans are now being widely used for the surveillance of patients having undergone curative resection for the primary colorectal cancer . Whole-body PET scanning in the patient with recurrent colorectal cancer has been reported to be more sensitive and accurate than Computed-Tomography (CT) and Magnetic-Resonance-Imaging (MRI). Moreover, PET is purported to be capable of differentiating among recurrent malignancy, scar, fibrosis, and necrosis, thus preventing the patients from futile surgery.15 With the above-mentioned reasons in mind, we then conducted this retrospective study to look at the efficacy of PET scan for directing surgery in patients with LRRCRC. We hypothesized that with the better diagnostic sensitivity and specificity, as compared to the conventional imaging methods (CT/MRI) in detecting recurrences of colorectal cancer, PET can positively affect the surgical decision-making and thus improve the treatment outcomes for patients with LRRCRCs.

ELIGIBILITY:
Inclusion Criteria:

i. patients with primary colorectal cancers undergoing R0 resection ii. Patients with final histopathologic reports documenting the pathologic Tumor-Node-Metastasis (pTNM) stage I, II, or III

Exclusion Criteria:

i. Patients with pTNM stage IV primary colorectal cancer ii. Patients with R1/2 resection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: These patients were further grouped into PET-driven vs CT/MRI/PET-driven vs non-surgery group
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
5-year overall survival | 10 year
  5-year overall survival

SECONDARY OUTCOMES:
Life expectancy | 10 year
  Median survival
Type of resection | 10 year
  Sham operation vs R0 vs R1 vs R2
Blood loss | 10 year
  recorded in mL
Operation time | 10 year
  recorded in minute
Type of surgical complication | 10 year
  specific complications; Clavien-Dindo classification
Hospitalization | 10 year
  recorded in day
Readmission | 10 year
  within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung LIANG, MD,PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan